CLINICAL TRIAL: NCT06247280
Title: Multicenter Prospective and Retrospective Cohort Study in Non-small Cell Lung Cancer Patients with EGFR Mutation: Korean EGFR Registry
Brief Title: Korean Registry of Non-Small Cell Lung Cancer Patients with EGFR Mutation
Status: Active, not recruiting | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Collaborators: The Korean Academy of Tuberculosis and Respiratory Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: YMC048
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Korean Registry of Non-Small Cell Lung Cancer Patients with EGFR mutation to collect and analyze the patient's clinical features, diagnosis, and treatment results.

DETAILED DESCRIPTION:
The Korean EGFR Registry is a prospective multicenter observational cohort study designed to enroll all stage EGFR-mutated non-small cell lung cancer (NSCLC) patients. However, due to the extended follow-up period required to confirm clinical outcomes, a retrospective cohort has been included. This retrospective cohort comprises patients with recurrent or metastatic NSCLC who began taking EGFR TKI after January 2021. The recruitment phase was planned to span 36 months, commencing in May 2022, with scheduled follow-up activities continuing until December 2026. The target enrollment for this study is set at 2,000 patients, with competitive enrollment to be carried out across 40 university hospitals in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 20-year-old with Korean nationality
2. A person who voluntarily signed the informed consent form for this study
3. All stage Non small cell lung cancer patients with EGFR mutation or Metastatic or recurred EGFR mutated NSCLC patients started with EGFR TKI treatment from 2021-01-01.

Exclusion Criteria:

1. A person who is not confirmed NSCLC histologically or cytologically.
2. A person who doesn't consent to the study.
3. A person who is unable to complete the study judged by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer of any stage with an EGFR mutation newly diagnosed after the date of IRB approval, or patients who started EGFR-targeted therapy for the first time after 2021-01-01 with metastatic or recurrent EGFR mutation non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2001 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of NSCLC patients with EGFR mutation | 12months, 18months, 24months, 36months
  Analysis of clinical characteristics and clinical outcomes in NSCLC patients with EGFR mutation
Clinical outcome of NSCLS patients with EGFR mutation | 12months, 18months, 24months, 36months
  Analysis of clinical characteristics and clinical outcomes in NSCLC patients with EGFR mutation
PFS | 12months, 18months, 24months, 36months
  PFS underwent palliative therapy according to stages in NSCLC patients with EGFR mutation
DFS | 12months, 18months, 24months, 36months
  DFS in patients underwent definitive therapy according to stages in NSCLC patients with EGFR mutation

SECONDARY OUTCOMES:
Diagnosis Test Method | up to 36months
  Frequency of diagnostic test methods according various clinical samples
Diagnosis Test Method | up to 36months
  Proportion of diagnostic test methods according various clinical samples
OS(Overall survival) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
ORR(overall response rate) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
DoR (duration of response) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
DCR (disease control rate) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
TTF (time to treatment failure) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
TTNF (time to next treatment) | up to 36months
  Exploration of clinical outcomes according to treatment modality in NSCLC patients with EGFR mutation
Analysis of metastatic sites and treatment patterns (especially brain and bone metastasis) | up to 36months
  Exploration of clinical characteristics and metastatic patterns in NSCLC patients with EGFR mutation
Adverse event profiles | up to 36months
  Adverse event profiles after lazertinib administration

CONTACTS AND LOCATIONS:
Overall Officials: Sae Young Lee, Study Director — Yuhan Corporation
Locations (39):
- South Korea (39):
  - Kyungpook National University Chilgok Hospital, Chilgok, Daegu
  - Hallym Univ. Medical Center. Chuncheon, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - The Catholic Univ. of Korea Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggido
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Catholic Yeouido Sungmo Hospital, Seoul, Seoul
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Samsung Changwon Hospital, Busan
  - Changwon Gyeongsang National University Hospital, Changwon
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang Univ. Hospital, Daejeon
  - Cheonnam National University Hwasun Hospital, Hwasun
  - Inha University Hospital, Incheon
  - The Catholic University of Korea Incheon St.Mary's Hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - The Catholic University Of Korea Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, University of Ulsan, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym UNIV. Medical Center, Seoul
  - Hanyang University Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Konkuk unversity hospital, Seoul
  - Kyunghee university hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: Undecided